CLINICAL TRIAL: NCT06991868
Title: A Multicenter Prospective Cohort Study on Monitoring Recurrence of Urothelial Carcinoma Based on Detection of Urinary Microscopic Residual Disease (MRD)
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UCMRD-010
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: NMIBC; MIBC; UTUC
Keywords: high-risk upper tract urothelial carcinoma (UTUC) (pT3-4 or N+); non-muscle invasive bladder cancer (NMIBC) (including low-risk, intermediate-risk, and high-risk/very-high-risk); muscle-invasive bladder cancer (MIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort I: 1. patients ≥18 years of age with full civil capacity at the time of signing the informed consent form;
  2. patients who provide a urine sample for MRD testing at the time of undergoing postoperative review;
  3. Pathologic type: required to be a pathologically confirmed uroepithelial tumor with a predominantly urothelial tumor with a primary site in the upper urinary tract (including the renal pelvis and ureters), and permitted to contain no more than 50% squamous differentiation, adenomatous differentiation, or sarcomatoid differentiation and are pT3/4 or any TpN+.
- Cohort II: 1. patients aged ≥18 years at the time of signing the informed consent form with full civil capacity;
  2. patients who provided a urine sample for central testing when they underwent postoperative review;
  3. Pathological type: a pathologically confirmed predominantly uroepithelial tumor with a primary site in the bladder is required, and is permitted to contain no more than 50% squamous differentiation, or adenoidal differentiation carcinoma in situ is permitted to be present or only in situ and the pathologic stage may be T1, Ta, or Tis (Cis).
- Cohort III: 1. patients aged ≥18 years at the time of signing the informed consent form with full civil capacity;
  2. patients providing urine samples for centralized testing prior to each cycle of treatment during neoadjuvant therapy;
  3. pathology type: a predominantly urothelial tumor with a TUR surgical pathology primary site in the bladder is required, and is permitted to contain no more than 50% squamous, adenomatous, or sarcomatoid differentiation (iii) Patients with pathologic stage T2 or MIBC on comprehensive imaging despite pathologic stage T1;
  4. Radical cystectomy after neoadjuvant therapy, including bladder, prostate, and seminal vesicles in men and bladder and uterus in women;
  5. lymph node dissection at least to the extent of the standard dissection for bladder cancer (including the area of the common iliac arteries below the bifurcation of the iliac arteries bilaterally and the area between the ipsoas and genitofemoral nerve to the ureter)
- Cohort IV: 1. patients aged ≥18 years at the time of signing the informed consent form with full civil capacity;
  2. patients to provide a urine sample for centralized testing at each review visit;
  3. pathology type: the TUR surgical pathology is required to be a predominantly uroepithelial tumor with a primary site in the bladder, and is allowed to contain no more than 50% squamous, adenomatous, or sarcomatous differentiation;
  4. there should be a centralized imaging to assess a clinical assessment of MIBC prior to TMT treatment;
  5. patients assessed as clinically CR after undergoing TMT who can continue to retain their bladder and do not require salvage cystotomy.

SUMMARY:
This was a multicenter, prospective, non-interventional, observational cohort study, and the enrolled patients were divided into four cohorts: cohort I was patients with high-risk upper tract urothelial carcinoma (UTUC) (pT3-4 or N+); cohort II was patients with non-muscle invasive bladder cancer (NMIBC) (including low-risk, intermediate-risk, and high-risk/very-high-risk); cohort III was patients with muscle-invasive bladder cancer (MIBC) to receive neoadjuvant therapy; and cohort IV was patients evaluated for complete response (CR) after standard trimodality therapy (TMT) treatment (i.e. patients with successful bladder preservation). Primary Objectives Cohorts I and IV: MRD score to assess the sensitivity and specificity of imaging recurrence/metastasis; Cohort II: MRD score to assess the sensitivity and specificity of tumor recurrence; Cohort III: MRD score to assess the sensitivity and specificity of tumor remnants. Secondary Objectives Cohorts I and IV: MRD score to assess the sensitivity and specificity of imaging recurrence subgroup and metastasis subgroup; Cohort II: MRD score to assess the sensitivity and specificity of different grades and stages of recurrent tumors; Cohort III: MRD scores to assess the sensitivity and specificity of different grades and stages of residual tumors.

ELIGIBILITY:
Cohort I:

Inclusion Criteria:

* patients ≥18 years of age with full civil capacity at the time of signing the informed consent form;
* patients who provide a urine sample for MRD testing at the time of undergoing postoperative review;
* Pathologic type: required to be a pathologically confirmed uroepithelial tumor with a predominantly urothelial tumor with a primary site in the upper urinary tract (including the renal pelvis and ureters), and permitted to contain no more than 50% squamous differentiation, adenomatous differentiation, or sarcomatoid differentiation and are pT3/4 or any TpN+.

Exclusion Criteria:

* Pathology after radical surgery that does not meet the criteria for enrollment;
* Predictable inability to meet the criteria for regular review at our center within 1 year postoperatively;
* Disagreement with regular cystoscopy and/or imaging (at least completion of one of CT or MR or PET/CT, with intervals between reviews as well as the specific items to be determined by the clinician);
* Already definite recurrence or metastasis;
* Concomitant combination of other active malignant neoplastic disease or a history of other malignant neoplastic disease within 5 years (excluding basal cell carcinoma and cervical carcinoma in situ after active treatment)

Cohort II:

Inclusion Criteria:

* patients aged ≥18 years at the time of signing the informed consent form with full civil capacity;
* patients who provided a urine sample for central testing when they underwent postoperative review;
* Pathological type: a pathologically confirmed predominantly uroepithelial tumor with a primary site in the bladder is required, and is permitted to contain no more than 50% squamous differentiation, or adenoidal differentiation carcinoma in situ is permitted to be present or only in situ and the pathologic stage may be T1, Ta, or Tis (Cis)

Exclusion Criteria:

* TUR pathology that does not meet the enrollment criteria;
* predictable inability to meet the regular review at our center within 1 year postoperatively;
* disagreement with regular cystoscopy and/or imaging (the content and type of imaging will be determined by the clinician);
* definite recurrence or metastasis already exists;
* concurrent combination of other active malignant neoplastic disease or a 5-year history of other malignant neoplastic disease history (excluding basal cell carcinoma and cervical carcinoma in situ after active treatment)

Cohort III:

Inclusion Criteria:

* patients aged ≥18 years at the time of signing the informed consent form with full civil capacity;
* patients providing urine samples for centralized testing prior to each cycle of treatment during neoadjuvant therapy;
* pathology type: a predominantly uroepithelial tumor with a TUR surgical pathology primary site in the bladder is required, and is permitted to contain no more than 50% squamous, adenomatous, or sarcomatoid differentiation (iii) Patients with pathologic stage T2 or MIBC on comprehensive imaging despite pathologic stage T1;
* Radical cystectomy after neoadjuvant therapy, including bladder, prostate, and seminal vesicles in men and bladder and uterus in women;
* lymph node dissection at least to the extent of the standard dissection for bladder cancer (including the area of the common iliac arteries below the bifurcation of the iliac arteries bilaterally and the area between the ipsoas and genitofemoral nerve to the ureter);
* the presence of evaluable lesions on imaging based on RECIST 1.1 criteria prior to neoadjuvant therapy.

Exclusion Criteria:

* TUR pathology that does not meet enrollment criteria;
* does not undergo radical total cystectomy or standard surgical scope;
* receives less than 2 cycles of neoadjuvant therapy;
* does not undergo regular imaging evaluations during preoperative neoadjuvant therapy;
* has no evaluable lesions prior to neoadjuvant therapy;
* already has definitively present distant metastases;
* concurrently combines other active malignant neoplastic disease or a history of other malignant neoplastic disease within 5 years (excluding basal cell carcinoma and cervical carcinoma in situ after active treatment).

Cohort IV:

Inclusion Criteria:

* patients aged ≥18 years at the time of signing the informed consent form with full civil capacity;
* patients to provide a urine sample for centralized testing at each review visit;
* pathology type: the TUR surgical pathology is required to be a predominantly urothelial tumor with a primary site in the bladder, and is allowed to contain no more than 50% squamous, adenomatous, or sarcomatous differentiation;
* there should be a centralized imaging to assess a clinical assessment of MIBC prior to TMT treatment;
* patients assessed as clinically CR after undergoing TMT who can continue to retain their bladder and do not require salvage cystotomy.

Exclusion Criteria:

* TUR pathology that does not meet the inclusion criteria;
* predictable inability to meet the regular review at our center within 1 year after surgery;
* no pre-treatment imaging at our center;
* disagreement with regularity of receiving imaging (the clinician decides on the content and type of imaging);
* residual lesions or metastases that are already clearly present;
* concurrent combination of other active malignant neoplastic diseases or a history of other malignant neoplastic diseases within 5 year history of other malignant neoplastic disease (excluding basal cell carcinoma and cervical carcinoma in situ after active treatment).

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with high-risk upper tract urothelial carcinoma (UTUC) (pT3-4 or N+), non-muscle invasive bladder cancer (NMIBC) (including low-risk, intermediate-risk, and high-risk/very-high-risk), and muscle-invasive bladder cancer (MIBC)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
UC MRD score | Cohort I: At begin of Cycle 1 and end of Cycle 6 (each cycle 21 days); Cohort II: every 6 months after surgery until 12 months; Cohort III: Baseline and The first day of thest neoadjuvant ther Cohort IV: every 6 months after TMT therapy until 12 months
  Provide 100 ml of morning urine for UC MRD testing at the appropriate collection node; assessment results were recorded as a score (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China